CLINICAL TRIAL: NCT06282653
Title: Postural and Muscle Fatigue Analysis of Endodontic Residents: A Research Proposal
Brief Title: Postural and Muscle Fatigue Analysis of Endodontic Residents
Status: Recruiting | Type: Observational
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Díaz-Flores García, Principal Investigator, Universidad Europea de Madrid
Other Study IDs: Endo-ergonomics
Record Dates: First submitted 2024-02-02; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Musculoskeletal System Disease; Position Sense Disorders; Symptoms and Signs; Postural; Defect; Endodontic Disease
Keywords: Endodontics; Musculoskeletal System; Ergonomics
MeSH Terms: conditions — Musculoskeletal Diseases; Somatosensory Disorders; Signs and Symptoms; Dental Pulp Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: 1st Year Students
- Group 2: 2nd year students

SUMMARY:
Musculoskeletal disorders (MSDs) are a significant occupational health problem for dentists and have been linked to a decline in quality of life, often leading to stress-related illnesses and early retirement. Poor posture, poor movement or imbalances in the neck or shoulders can lead to the three most common pain syndromes in dentistry. The objectives of this study were to evaluate the working position adopted during an endodontic procedure and to determine the perception of symptoms of musculoskeletal disorders in first and second year students of the Master in Advanced Endodontics at the European University of Madrid (UEM), using the standardised Nordic Kuorinka questionnaire supplemented by a form with socio-demographic variables. This study has a descriptive cross-sectional observational design and included 10 students selected by convenience sampling. A video camera was used to record the procedures from three different angles for a maximum of 5 minutes. The information was processed using Microsoft Excel spreadsheet software, and the video recordings were assessed using Rodgers' Muscular Fatigue Analysis (RMFA) and Rapid Upper Limb Assessment (RULA).

DETAILED DESCRIPTION:
The unit of analysis for this study consisted of the first and second year students of the Master's in Endodontics programme at the European University of Madrid (UEM) who completed the two years of annual clinical practice during the years 2022/24. A total of 10 students were enrolled over the two years of training, treating 30 patients (3 patients per student) in the first year and another 30 patients in the second year (for a total of 22 months). A video camera was used to record the procedures from three different angles for a maximum of 5 minutes (two side views - right and left - and one frontal view) on different patients, following the National Institute for Occupational Safety and Health (NIOSH) Protocol for Video Recording for Job Analysis and Risk Assessment. The selected endodontic procedure focused exclusively on upper or lower first molars during the opening and ultrasonic search for the fourth canal in upper first molars or the search for the mesiobuccal canal in lower first molars. The standardised Nordic Kuorinka Musculoskeletal Symptom Perception Questionnaire was used as the measuring instrument. Questionnaire data were collected using a spreadsheet program (Microsoft Excel).

ELIGIBILITY:
Inclusion Criteria:

- Students of the Master's Degree in Endodontics of the European University of Madrid (UEM), who have completed the two years of the annual teaching period of clinical practice.

Exclusion Criteria:

* Subjects previously diagnosed with a musculoskeletal disorder.
* Subjects who had suffered previous trauma affecting the musculoskeletal system.
* Pregnant women in their third trimester.
* Subjects who refused to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1st and 2nd year students of the Master's Degree in Endodontics of the European University of Madrid (UEM), who have completed the two years of the annual teaching period of clinical practice during the years 2022/24.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Symptom Perception | January 2023 - July 2024
  The standardized Nordic Kuorinka Musculoskeletal Symptom Perception Questionnaire will be used as a measurement instrument. Data from the questionnaires will be compiled in a spreadsheet program (Microsoft Excel); measures of central tendency and dispersion will be calculated as well as tables and figures. Sociodemographic variables such as age, sex, grade, weight, height, symptoms of musculoskeletal disorders, body regions affected and times of symptom onset will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Perez Alfayate, PHD, Study Chair — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
The data obtained will be used for scientific publications.

REFERENCES:
- [Result] Zarra T, Lambrianidis T. Musculoskeletal disorders amongst Greek endodontists: a national questionnaire survey. Int Endod J. 2014 Aug;47(8):791-801. doi: 10.1111/iej.12219. Epub 2014 Jan 11. PMID 24283200
- [Result] Hayes M, Cockrell D, Smith DR. A systematic review of musculoskeletal disorders among dental professionals. Int J Dent Hyg. 2009 Aug;7(3):159-65. doi: 10.1111/j.1601-5037.2009.00395.x. PMID 19659711
- [Result] McAtamney L, Nigel Corlett E. RULA: a survey method for the investigation of work-related upper limb disorders. Appl Ergon. 1993 Apr;24(2):91-9. doi: 10.1016/0003-6870(93)90080-s. PMID 15676903

DOCUMENTS (2):
  • Study Protocol (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT06282653/Prot_000.pdf
  • Informed Consent Form (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT06282653/ICF_001.pdf